CLINICAL TRIAL: NCT04711460
Title: Mindfulness, Group Therapy and Psychosis; Training Decreases Anxiety and Depression in Outpatients With a Psychotic Disorder in a Non-Randomized Within Group Comparison
Brief Title: Mindfulness, Group Therapy and Psychosis; Training Decreases Anxiety and Depression
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00005035
Record Dates: First submitted 2020-12-15; First posted 2021-01-15 (Actual); Results first posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2023-05

CONDITIONS: Psychosis
Keywords: mindfulness; group therapy
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Younger participants: Participants were adults ages19 to 29 years who recieved CBT and 10 minutes of Mindfulness Training and practice in group therapy.
  Interventions: Behavioral: Younger participants
- Older participants: Participants were adults ages 30-54 years who received CBT and 10 minutes of Mindfulness Training and practice in group therapy.
  Interventions: Behavioral: Older participants
- Treatment As Usual (TAU): . Participants in the "Treatment As Usual" (TAU) group had Cognitive Behavioral Therapy and education about the mindfulness process, but no practice of the mindfulness technique as a group.
  Interventions: Behavioral: TAU
- TAU plus mindfulness practice: Participants in the TAU plus Mindfulness Practice had Cognitive Behavioral Therapy (CBT) and 10 minutes of mindfulness practice in group therapy sessions.
  Interventions: Behavioral: TAU + MIndfulness practice

INTERVENTIONS:
Behavioral: Younger participants — Younger Participants 19-29 years received TAU + Tx over 5 weeks
  Groups: Younger participants
Behavioral: Older participants — older participants 30-54 years received TAU + Tx over 5 weeks
  Groups: Older participants
Behavioral: TAU — Participants received TAU or Treatment As Ususal, Cognitive Behavior Therapy only
  Groups: Treatment As Usual (TAU)
Behavioral: TAU + MIndfulness practice — Participants received TAU + mindfulness training
  Groups: TAU plus mindfulness practice

SUMMARY:
The objective of this non-randomized, within-group comparison was to evaluate the addition of mindfulness as a new technique in an outpatient group therapy program for participants diagnosed with a psychotic spectrum disorder, alongside of cognitive behavioral therapy.

DETAILED DESCRIPTION:
Participants completed the Patient Health Questionnaire-9 (PHQ-9), and the Generalized Anxiety Disorder 7-item scale (GAD-7), at admission and discharge. The first experiment compared scores of those who received mindfulness training plus standard psychiatric treatment or treatment as usual (TAU) against those who received TAU. The second experiment compared age using matched scores from participants who received mindfulness training plus TAU. Participants attended group therapy for a five-week minimum, and were taught the mindfulness practices of breath, acceptance, observation, remaining non-judgmental, and letting go.

ELIGIBILITY:
Inclusion Criteria:

* All Diagnostic Statistical Manual, Fifth edition, (DSM-5) diagnoses that included a psychosis spectrum disorder

Exclusion Criteria:

* those lacking symptoms of psychosis

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: . Eligible participants had a
  DSM-5 diagnosis which included: 295.2 Schizophrenia, Catatonia type, 295.3 Schizophrenia, Paranoid Type, 295.4 Schizophreniform Disorder, 295.70 Schizoaffective Disorder, Depressed Type or Bipolar Type, 295.9 Schizophrenia, Unspecified, 296.34 Major Depressive Disorder, With Psychotic Features, 296.54 Bipolar Disorder, With Psychotic Features, 297.1 Delusional Disorder, 298.8 Brief Psychotic Disorder, 298.9 Unspecified Schizophrenia and Other Psychotic Disorders, 301.22 Schizotypal Personality Disorder.
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joan D Lund, Psy.D., Principal Investigator — University of Minnesota

IPD SHARING:
Plan to Share IPD: No
Data is not available for sharing

REFERENCES:
- [Background] Brown KW, Ryan RM. The benefits of being present: mindfulness and its role in psychological well-being. J Pers Soc Psychol. 2003 Apr;84(4):822-48. doi: 10.1037/0022-3514.84.4.822. PMID 12703651
- [Background] Brown RL, Rounds LA. Conjoint screening questionnaires for alcohol and other drug abuse: criterion validity in a primary care practice. Wis Med J. 1995;94(3):135-40. PMID 7778330
- [Background] Chadwick P, Hughes S, Russell D, Russell I, Dagnan D. Mindfulness groups for distressing voices and paranoia: a replication and randomized feasibility trial. Behav Cogn Psychother. 2009 Jul;37(4):403-12. doi: 10.1017/S1352465809990166. Epub 2009 Jun 23. PMID 19545481
- [Background] Chadwick P. Mindfulness for psychosis. Br J Psychiatry. 2014;204:333-4. doi: 10.1192/bjp.bp.113.136044. PMID 24785766
- [Background] Chadwick P, Strauss C, Jones AM, Kingdon D, Ellett L, Dannahy L, Hayward M. Group mindfulness-based intervention for distressing voices: A pragmatic randomised controlled trial. Schizophr Res. 2016 Aug;175(1-3):168-173. doi: 10.1016/j.schres.2016.04.001. Epub 2016 Apr 14. PMID 27146475
- [Background] Chadwick P. Mindfulness for psychosis: a humanising therapeutic process. Curr Opin Psychol. 2019 Aug;28:317-320. doi: 10.1016/j.copsyc.2019.07.022. Epub 2019 Jul 18. PMID 31382104
- [Background] Chien WT, Thompson DR. Effects of a mindfulness-based psychoeducation programme for Chinese patients with schizophrenia: 2-year follow-up. Br J Psychiatry. 2014 Jul;205(1):52-9. doi: 10.1192/bjp.bp.113.134635. Epub 2014 May 8. PMID 24809397
- [Background] Dhalla S, Kopec JA. The CAGE questionnaire for alcohol misuse: a review of reliability and validity studies. Clin Invest Med. 2007;30(1):33-41. doi: 10.25011/cim.v30i1.447. PMID 17716538
- [Background] Dixon LB, Holoshitz Y, Nossel I. Treatment engagement of individuals experiencing mental illness: review and update. World Psychiatry. 2016 Feb;15(1):13-20. doi: 10.1002/wps.20306. PMID 26833597
- [Background] Ellett L. Mindfulness for paranoid beliefs: evidence from two case studies. Behav Cogn Psychother. 2013 Mar;41(2):238-42. doi: 10.1017/S1352465812000586. Epub 2012 Sep 14. PMID 22974494
- [Background] Hayes SC. Acceptance and Commitment Therapy, Relational Frame Theory, and the Third Wave of Behavioral and Cognitive Therapies - Republished Article. Behav Ther. 2016 Nov;47(6):869-885. doi: 10.1016/j.beth.2016.11.006. Epub 2016 Nov 10. PMID 27993338
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Khoury B, Lecomte T, Gaudiano BA, Paquin K. Mindfulness interventions for psychosis: a meta-analysis. Schizophr Res. 2013 Oct;150(1):176-84. doi: 10.1016/j.schres.2013.07.055. Epub 2013 Aug 15. PMID 23954146
- [Background] Langer AI, Cangas AJ, Salcedo E, Fuentes B. Applying mindfulness therapy in a group of psychotic individuals: a controlled study. Behav Cogn Psychother. 2012 Jan;40(1):105-9. doi: 10.1017/S1352465811000464. Epub 2011 Sep 9. PMID 21902854
- [Background] Morrison AP, Wells A. A comparison of metacognitions in patients with hallucinations, delusions, panic disorder, and non-patient controls. Behav Res Ther. 2003 Feb;41(2):251-6. doi: 10.1016/s0005-7967(02)00095-5. PMID 12547384
- [Background] Mundt JC, Greist JH, Jefferson JW, Federico M, Mann JJ, Posner K. Prediction of suicidal behavior in clinical research by lifetime suicidal ideation and behavior ascertained by the electronic Columbia-Suicide Severity Rating Scale. J Clin Psychiatry. 2013 Sep;74(9):887-93. doi: 10.4088/JCP.13m08398. PMID 24107762
- [Background] Posner K, Brown GK, Stanley B, Brent DA, Yershova KV, Oquendo MA, Currier GW, Melvin GA, Greenhill L, Shen S, Mann JJ. The Columbia-Suicide Severity Rating Scale: initial validity and internal consistency findings from three multisite studies with adolescents and adults. Am J Psychiatry. 2011 Dec;168(12):1266-77. doi: 10.1176/appi.ajp.2011.10111704. PMID 22193671
- [Background] Ratcliffe M, Wilkinson S. How anxiety induces verbal hallucinations. Conscious Cogn. 2016 Jan;39:48-58. doi: 10.1016/j.concog.2015.11.009. Epub 2015 Dec 9. PMID 26683229
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Terrill AL, Hartoonian N, Beier M, Salem R, Alschuler K. The 7-item generalized anxiety disorder scale as a tool for measuring generalized anxiety in multiple sclerosis. Int J MS Care. 2015 Mar-Apr;17(2):49-56. doi: 10.7224/1537-2073.2014-008. PMID 25892974
- [Result] Birchwood M, Chadwick P. The omnipotence of voices: testing the validity of a cognitive model. Psychol Med. 1997 Nov;27(6):1345-53. doi: 10.1017/s0033291797005552. PMID 9403906
- [Result] Bach P, Hayes SC. The use of acceptance and commitment therapy to prevent the rehospitalization of psychotic patients: a randomized controlled trial. J Consult Clin Psychol. 2002 Oct;70(5):1129-39. doi: 10.1037//0022-006x.70.5.1129. PMID 12362963
- [Result] Baer RA, Smith GT, Lykins E, Button D, Krietemeyer J, Sauer S, Walsh E, Duggan D, Williams JM. Construct validity of the five facet mindfulness questionnaire in meditating and nonmeditating samples. Assessment. 2008 Sep;15(3):329-42. doi: 10.1177/1073191107313003. Epub 2008 Feb 29. PMID 18310597

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There was no recruitment used for this study.
Pre-assignment Details: All participants assessed and enrolled had a DSM-V diagnosis that included psychosis. They participated twice a week for 5 weeks.
  Pre/post-test scores were collected and compared.
Groups:
- 1: TAU: 1: The Treatment as usual (TAU) group received only Cognitive Behavioral Therapy (CBT)
- The TAU + Treatment Group: The TAU plus Mindfulness Training received CBT and Mindfulness Training
- Younger Participants: scores were compared on pre/post-test scores
- Older Participants: pre/post-test scores were compared
Period: Overall Study
Arm/Group | 1: TAU | The TAU + Treatment Group | Younger Participants | Older Participants
Started | 32 | 32 | 26 | 26
Completed | 32 | 32 | 26 | 26
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The number of participants in each study: Treatment as usual (TAU) versus TAU + Mindfulness and the Younger versus Older study.
Groups:
- Treatment as Usual CBT: Treatment as usual (TAU group) Participants in the "Treatment as usual" (TAU) group had Cognitive Behavioral Therapy only.
- Treatment as Usual + Mindfulness Training: (TAU + TX group) Participants had Cognitive Behavioral Therapy (CBT), mindfulness training
- Younger Participants: Younger participants pre/post test scores were compared
- Older Participants: Older participants pre/post test scores were compared
- Total: Total of all reporting groups
Arm/Group | Treatment as Usual CBT | Treatment as Usual + Mindfulness Training | Younger Participants | Older Participants | Total
Number analyzed (Participants) | 32 | 32 | 26 | 26 | 116
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 32 | 32 | 26 | 26 | 116
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex/Gender, Customized [Number; unit: participants] — Categories for gender include Male, Female, and Transgender. Participants were counted in each category. Population: Gender is defined as male, female, and transgender for each category
  participants
    Male | 19 | 13 | 10 | 11 | 53
    Female | 9 | 13 | 6 | 11 | 39
    Transgender | 4 | 6 | 10 | 4 | 24
Race/Ethnicity, Customized [Number; unit: participants] — The number of participants in each ethnic category were counted.
  participants
    Ethnicity: Caucasian | 20 | 15 | 10 | 13 | 58
    Ethnicity: African American | 5 | 7 | 6 | 4 | 22
    Ethnicity: Native American | 3 | 5 | 6 | 3 | 17
    Ethnicity: Hispanic | 1 | 0 | 2 | 1 | 4
    Ethnicity: Asian | 0 | 2 | 0 | 5 | 7
    Ethnicity: Jewish | 1 | 3 | 1 | 0 | 5
    Ethnicity: African continent | 2 | 0 | 1 | 0 | 3
Region of Enrollment [Number; unit: participants] — Participants were enrolled in an Outpatient Mental Health program in Minneapolis, Minnesota, USA.
  participants
    United States | 32 | 32 | 26 | 26 | 116
PHQ-9 and GAD-7 Number of Participants [Mean (Standard Deviation); unit: units on a scale]
  PHQ-9 Scores: Mean (Standard Deviation) Unit of measures: scores on a scale | 9.32 (6.4) | 12.31 (7.19) | 11.84 (5.9) | 12.34 (6.9) | 11.45 (6.15)
  GAD-7 Scores: Mean (Standard Deviation) Unit of measures: scores on a scale | 6.25 (5.4) | 10.09 (5.59) | 9.15 (5.39) | 11.42 (5.13) | 9.23 (5.38)

OUTCOME MEASURES:

1. Primary Outcome: Change in Generalized Anxiety Disorder-7 Pre/Post Test at Week 5
Description: The Generalized Anxiety Disorder 7-item scale (GAD-7) is a 7-item survey of how often patients are bothered by symptoms of anxiety. Items are rated from 0 (not at all) to 3 (nearly every day). The total score is a sum of item scores and ranges from 0 (minimal depression) to 27 (severe depression). Outcome is reported as the change from baseline to approximately 5 weeks.
  Pre / Post-test scores were compared.
Time Frame: Five weeks
Population: The Generalized Anxiety Disorder 7 number of participants for two studies: Treatment as usual vs TAU + Mindfulness study and the Younger versus older study.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Treatment as Usual: The Treatment as usual (TAU) group received only Cognitive Behavioral Therapy (CBT)
- TAU + Mindfulness Training: The TAU plus Mindfulness Training received CBT and Mindfulness Training.
- Younger Participants; Older Participants: Pre/post test scores were obtained from younger participants who received TAU + Mindfulness Training
Arm/Group | Treatment as Usual | TAU + Mindfulness Training | Younger Participants | Older Participants
Number analyzed (Participants) | 32 | 32 | 26 | 26
units on a scale | 4.68 (5.4) | 6.28 (5.59) | 3.96 (5.39) | 7.38 (5.13)
Statistical Analysis 1: Comparison: Treatment as Usual vs TAU + Mindfulness Training; Test type: Superiority — Threshold of statistically significance was set at p=0.05. No power calculation was conducted; p = 0.003, t-test, 2 sided — Threshold of statistically significance was set at p=0.05. No power calculation was conducted; Threshold of statistically significance was set at p=0.05. No power calculation was conducted; Mean Difference (Final Values) = 0.003, Standard Deviation 5.59
Statistical Analysis 2: Comparison: Treatment as Usual vs TAU + Mindfulness Training; Test type: Superiority — The threshold for statistical significance was set at p=0.05. No power analysis was conducted; p = 0.009, ANOVA — Threshold of statistically significance was set at p=0.05. No power calculation was conducted; Threshold of statistically significance was set at p=0.05. No power calculation was conducted; Mean Difference (Final Values) = 0.009, Standard Deviation 5.59 — Threshold of statistically significance was set at p=0.05. No power calculation was conducted
Statistical Analysis 3: Comparison: Treatment as Usual vs TAU + Mindfulness Training; Test type: Superiority — The Tukey Kramer Post Hoc Test q value = 0.05 threshold; p < 0.05, Tukey Kramer Post-Hoc — Threshold of statistically significance was set at p=0.05. No power calculation was conducted; Threshold of statistically significance was set at p=0.05; Mean Difference (Final Values) = 0.05, Standard Error of Mean 0.609 — Threshold of statistically significance was set at p=0.05. No power calculation was conducted
Statistical Analysis 4: Comparison: Younger Participants vs Older Participants; Threshold of statistically significance was set at p=0.05. No power calculation was conducted; Test type: Superiority — Threshold of statistically significance was set at p=0.05. No power calculation was conducted; p = 0.003, t-test, 2 sided — Threshold of statistically significance was set at p=0.05. No power calculation was conducted; Threshold of statistically significance was set at p=0.05. No power calculation was conducted; Mean Difference (Final Values) = 0.05, Standard Deviation 5.13 — Threshold of statistically significance was set at p=0.05. No power calculation was conducted
Statistical Analysis 5: Comparison: Younger Participants vs Older Participants; Threshold of statistically significance was set at p=0.05. No power calculation was conducted; Test type: Superiority; p = 0.454, ANOVA — Threshold of statistically significance was set at p=0.05. No power calculation was conducted; Threshold of statistically significance was set at p=0.05. No power calculation was conducted; Mean Difference (Final Values) = 0.05, Standard Deviation 5.07 — Threshold of statistically significance was set at p=0.05. No power calculation was conducted

2. Primary Outcome: Change in Patient Health Questionnaire-9 Score From Pre / Post-test at Week 5
Description: The Patient Health Questionnaire (PHQ-9) is a 9-item survey of how often patients are bothered by symptoms of depression. Items are rated from 0 (not at all) to 3 (nearly every day). The total score is a sum of item scores and ranges from 0 (minimal depression) to 27 (severe depression). Outcome is reported as the change from baseline to approximately 5 weeks.
Time Frame: Five weeks
Population: The Patient Health Questionnaire-9 scale number of participants in each study: The Treatment as usual (TAU) versus TAU + Mindfulness and the Younger versus Older study.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Treatment as Usual: The Treatment as usual (TAU) group received Cognitive Behavioral Therapy (CBT) only. The TAU + Mindfulness Training group received CBT and Mindfulness Training and practiced it as a group.
- TAU + Mindfulness Training: The group received CBT and Mindfulness Training and practiced it as a group.
- Younger Participants: Younger participants received TAU + Mindfulness Training.
- Older Participants: Older participants received TAU + Mindfulness Training.
Arm/Group | Treatment as Usual | TAU + Mindfulness Training | Younger Participants | Older Participants
Number analyzed (Participants) | 32 | 32 | 26 | 26
units on a scale | 6.68 (6.4) | 6.96 (7.19) | 3.96 (5.39) | 7.38 (5.13)
Statistical Analysis 1: Comparison: Treatment as Usual vs TAU + Mindfulness Training; Test type: Superiority — Threshold of statistically significance was set at p=0.05. No power calculation was conducted; p = 0.002, t-test, 2 sided — Threshold of statistically significance was set at p=0.05. No power calculation was conducted; Threshold of statistically significance was set at p=0.05. No power calculation was conducted; Mean Difference (Final Values) = 0.05, Standard Deviation 7.194 — Threshold of statistically significance was set at p=0.05. No power calculation was conducted
Statistical Analysis 2: Comparison: Treatment as Usual vs TAU + Mindfulness Training; Threshold of statistically significance was set at p=0.05. No power calculation was conducted; Test type: Superiority; p = 0.054, ANOVA — Threshold of statistically significance was set at p=0.05. No power calculation was conducted; Threshold of statistically significance was set at p=0.05. No power calculation was conducted; Mean Difference (Final Values) = 0.05, Standard Deviation 6.09 — Threshold of statistically significance was set at p=0.05. No power calculation was conducted
Statistical Analysis 3: Comparison: Younger Participants vs Older Participants; Threshold of statistically significance was set at p=0.05. No power calculation was conducted; Test type: Superiority — Threshold of statistically significance was set at p=0.05. No power calculation was conducted; p = 0.019, t-test, 2 sided — Threshold of statistically significance was set at p=0.05. No power calculation was conducted; Threshold of statistically significance was set at p=0.05. No power calculation was conducted; Mean Difference (Final Values) = 0.05, Standard Deviation 6.93 — Threshold of statistically significance was set at p=0.05. No power calculation was conducted
Statistical Analysis 4: Comparison: Younger Participants vs Older Participants; Threshold of statistically significance was set at p=0.05. No power calculation was conducted; Test type: Superiority — Threshold of statistically significance was set at p=0.05. No power calculation was conducted; p = 0.101, ANOVA — Threshold of statistically significance was set at p=0.05. No power calculation was conducted; Threshold of statistically significance was set at p=0.05. No power calculation was conducted; Mean Difference (Final Values) = 0.05, Standard Deviation 6.04

3. Secondary Outcome: CAGE-Adapted to Include Drug Use (CAGE-AID)
Description: The Cut-Annoyed-Guilty-Eye (CAGE) adapted to include drug use (CAGE-AID) is a screening tool to assess drug use. Participants are asked to answer yes (score of 1) or no (score of 0) to 4 questions about their drug use. Scores range from 0 to 4 with higher scores indicating greater substance use disorder. A score of 2 or higher indicates a problem with alcohol or drugs and is clinically significant. Outcome is reported as the number of participants who scored 2 or lower.
Time Frame: baseline only
Population: The CAGE-AID was used to determine sobriety in all participants, and was done before admission to the program. Scores must be below 2 and indicate no problems with alcohol or drugs.
Measure: Count of Participants; unit: Participants
Groups:
- The Treatment as Usual (TAU) Group: The Treatment as usual (TAU) group received Cognitive Behavioral Therapy (CBT) only.
- TAU + Mindfulness Group: The TAU + Mindfulness group received Cognitive Behavioral Therapy (CBT) and Mindfulness Training and practiced it with the group.
Arm/Group | The Treatment as Usual (TAU) Group | TAU + Mindfulness Group | Younger Participants | Older Participants
Number analyzed (Participants) | 32 | 32 | 26 | 26
Participants | 32 | 32 | 26 | 26

4. Secondary Outcome: The Columbia Suicide Severity Rating Scale (C-SSRS)
Description: The Columbia Suicide Severity Rating Scale, or C-SSRS, measures four constructs: the severity of ideation, the intensity of ideation, behavior, and lethality. Items are rated on a scale from 0-4: Eligible participants scored at 2 or lower.
  1. Only one time
  2. A few times
  3. A lot
  4. All the time
  0) Don't know/Not applicable
  The Columbia was done prior to being considered for the Outpatient Mental Health program by another licensed mental health staff in another department. Only those who scored at 1-2 would be considered for Outpatient. Outcome is reported as the number of participants who score a one or two on the scale, which means they are considered safe to participate.
Time Frame: baseline only
Measure: Count of Participants; unit: Participants
Groups:
- 1: The TAU Group: 1: The Treatment as usual (TAU) group received only Cognitive Behavioral Therapy (CBT).
- The TAU + TX Group: The TAU plus Mindfulness Training received CBT and Mindfulness Training.
- Younger Participants Scores: Younger participants received TAU + mindfulness training.
Arm/Group | 1: The TAU Group | The TAU + TX Group | Younger Participants Scores | Older Participants
Number analyzed (Participants) | 32 | 32 | 26 | 26
Participants | 32 | 32 | 26 | 26

ADVERSE EVENTS:
Time Frame: Data was collected over two years to obtain results for the groups.
Description: Data was collected over two years to obtain results for the groups. All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed
Groups:
- 1: The TAU Group / TAU vs TAU + TX: The Treatment as usual (TAU) group received only Cognitive Behavioral Therapy (CBT) and did not practice the Mindfulness as a group.
- The TAU + TX Group / TAU vs TAU + TX: The TAU plus Mindfulness Training received CBT and Mindfulness Training, which included practice as a group
- Younger Participants / Younger vs Older Scores: Younger vs Older participant scores were compared on pre/post-test scores
- Older Participants / Younger vs Older Scores: Younger vs Older participant pre/post-test scores were compared
Arm/Group | 1: The TAU Group / TAU vs TAU + TX | The TAU + TX Group / TAU vs TAU + TX | Younger Participants / Younger vs Older Scores | Older Participants / Younger vs Older Scores
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32 | 0/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32 | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 0/32 | 0/32 | 0/26 | 0/26

LIMITATIONS AND CAVEATS:
Limitations and caveats include the sample size. If a larger data base was collected, more significant results may have occurred. Data collection assumes that all participants will answer honestly on both scales. The financial resources and equipment were limited to what the author provided, as there were no grants. The setting was a group room, and some participants may prefer to be outside or be alone.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-12): https://cdn.clinicaltrials.gov/large-docs/60/NCT04711460/Prot_SAP_000.pdf